CLINICAL TRIAL: NCT04513431
Title: A Study Evaluating the Safety and Preliminary Efficacy of Anti-CEA CAR-T Cells for the Prevention of Postoperative Recurrence and Metastasis of Stage III Colorectal Cancer or Liver Metastasis of Colorectal Cancer
Brief Title: A Clinical Research of CAR T Cells Targeting CEA Positive Colorectal Cancer (CRC)
Acronym: CRC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: HuaDao (Shanghai) Biomedical Co., Ltd. (Other)
Responsible Party: Principal Investigator, Mei Wang, Director of Oncology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RJBY_anti-CEA CAR-T_CRC01
Record Dates: First submitted 2020-07-31; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Stage III Colorectal Cancer; Colorectal Cancer Liver Metastasis
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colorectal cancer (Experimental): Colorectal cancer treated with T cells modified with Anti-CEA-CAR T.
  Interventions: Biological: Anti-CEA-CAR T

INTERVENTIONS:
Biological: Anti-CEA-CAR T — T cells modified with CEA targeted chimeric antigen receptor.

SUMMARY:
The main purpose of this research is to verify the safety of CEA targeted chimeric antigen receptor T cells and to determine the proper dosage of CAR T cells infused.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR)-modified T cells have demonstrated great successes in treating even late stage cluster of differentiation antigen 19 (CD19) positive B cell malignancies. But it has few studies in solid tumors. The carcino-embryonic antigen(CEA) is widely expressed in cancers like gastric cancer, lung cancer, pancreatic cancer, breast cancer and colorectal cancer. To confirm if CAR T cells still function in solid tumors, we have developed anti-CEA CAR-modified T cells. Preclinical studies have demonstrated effective killing of CEA target cells. In this study, the CEA CARs, will be evaluated in CEA positive gastric cancer. The primary goal is to confirm its adverse effects including cytokine storm response and any other adverse effects. In addition, tumor targeting and disease status after treatment will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. CEA positive T4/N2 high-risk stage-Ⅲ colorectal cancer after surgery or patients with colorectal cancer liver metastasis after R0 surgery;
2. Patients whose serum CEA ≥11 ng/mL;
3. Life expectancy ≥ 3 months;
4. PS score 0-2, KPS score ≥60;
5. >3 CTC/7.5 mL blood sample;
6. Patients who plan to use XELOX chemotherapy after surgery;
7. Patients must have adequate organ function , such as NYHA heart function classification grade III or higher, no severe anemia, hypoxia; liver function: total bilirubin ≤ 1.5 × ULN (total bilirubin ≤ 3 × ULN when liver metastasis), ALT≤2.5×ULN, AST≤2.5×ULN (ALT or/and AST≤5×ULN when liver metastasis); renal function: blood creatinine ≤1.5 × ULN and creatinine clearance ≥50 mL/min, only when blood creatinine ≤ Calculate the creatinine clearance rate when 1.5 × ULN;
8. Sufficient peripheral blood can be obtained through peripheral veins without contraindications to apheresis;
9. Patients of childbearing age have no birth plans and take effective contraceptive measures during the study period and within 1 year after the study.

Exclusion Criteria:

1. Patients who have a history of severe central nervous system disease;
2. Other organ metastases except liver;
3. Patients who have non malignant diseases, including autoimmune diseases, primary immunodeficiency diseases or obstructive or restrictive respiratory diseases;
4. Patients received car-t or other gene modified T cell therapy previously;
5. Patients who plan to use other targeted anti-tumor drugs;
6. Patients who participated in other clinical studies within 30 days before screening or planned to participate in other clinical studies during the study period;
7. Patients who have syphilis or HIV / HBV / HCV / HPV / EBV / CMV infection ; HBV-DNA copy number ≥ 1 × 10 ^ 5 copies / ml is required for HBV seropositive patients;
8. Patients who have uncontrollable systemic infectious diseases;
9. Patients who have multiple malignant tumor;
10. Patients who received or may need Chinese herbal medicine, systemic glucocorticoid or other immunosuppressants within 2 weeks before enrollment;
11. Patient who are pregnancy and lactating;
12. Patients who have severe gastroduodenal ulcer, ulcerative colitis and other intestinal inflammation;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-08-30 (Estimated); Primary Completion 2021-03-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events that related to treatment | 4 weeks
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)

SECONDARY OUTCOMES:
Survival time of Anti-CEA CAR T cells in vivo. | 3 months
  To evaluate the presence of circulating CAR T cells with flow cytometry and real time PCR in patient blood.
Efficacy of anti-CEA CAR T cells to confirm the ability of CAR T cells to kill CEA positive cancer cells | 6 months
  To evaluate the presence of circulating tumor cells with flow cytometry and real time PCR in patient blood.
Maximum tolerated dose (MTD) of CEA targeted CAR T cells | 4 weeks
  To confirm the maximum tolerated dose of CEA targeted CAR T cells.

CONTACTS AND LOCATIONS:
Overall Officials: Ren Zhao, Medical PhD, Principal Investigator — Ruijin Hospital; Mei Wang, Medical PhD, Principal Investigator — Ruijin Hospital; Chen xianze, Medical PhD, Study Chair — Ruijin Hospital; Liu Kun, Medical PhD, Study Chair — Ruijin Hospital; Shi Yiqing, Medical PhD, Study Chair — Ruijin Hospital; Wang Chen, Medical PhD, Study Chair — Ruijin Hospital; He Qianyun, Medical PhD, Study Chair — Ruijin Hospital; Mao Dongliang, Medical PhD, Study Chair — Ruijin Hospital

IPD SHARING:
Plan to Share IPD: No